CLINICAL TRIAL: NCT03221075
Title: CLARITY - Clinical Implications of Azole-Resistant Aspergillosis in Hematological Malignancy
Brief Title: Clinical Implications of Azole-Resistant Aspergillosis in Hematological Malignancy
Acronym: CLARITY
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Oliver A. Cornely, Prof., University Hospital of Cologne
Other Study IDs: 17-024
Record Dates: First submitted 2017-05-09; First posted 2017-07-18 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Invasive Aspergillosis
Keywords: Invasive Aspergillosis; Azole resistance; Aspergillus fumigatus; Efficacy of antifungal therapy; Patient registry
MeSH Terms: interventions — Registries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasive Aspergillosis
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — There is no intervention.

SUMMARY:
In order to determine the efficacy of antifungal therapy in patients with documented azole-resistant invasive Aspergillosis (IA), anonymized clinical information of patients with a hematological malignancy with a culture-positive invasive fungal infection caused by Aspergillus fumigatus are collected in an online registry. Respective fungal isolates are analysed for azole susceptibility and resistance mechanisms. Patients diagnosed with an IA in 2016 and later are included in the study.

DETAILED DESCRIPTION:
For mold-active azoles (e.g. isavuconazole, itraconazole, posaconazole and voriconazole), cross-resistance of Aspergillus spp. is an increasingly recognized problem. The study aims to determine the efficacy of antifungal therapy in patients with documented azole-resistant IA. On the basis of this study, it will be possible to assess the clinical implications of IA caused by azole-resistant versus azole-susceptible Aspergillus spp.

The investigators aim at collecting at least 55 azole-resistant and 130 azole-susceptible cases. Cases diagnosed with an IA by culture from January 1st, 2016 onwards with an underlying hematological malignancy are eligible for inclusion. Culture of azole-resistant cases must be provided for confirmation of the species, sequencing for azole-resistance mutations and determination of MIC using the EUCAST reference method. Isolates obtained from patients with presumed azole-susceptible disease will be analyzed to confirm the wild type phenotype.

Eligible azole-resistant and azole-susceptible IA cases will be documented using the web-based case report form. If there is ≥1 resistant isolate, the patient fulfills the definition of a resistant case. Patient level data will be recorded at the respective study centres in a continuous fashion. Data items to be documented will include: demographic data; type and status of underlying conditions; concurrent immunosuppressive treatment; diagnostic measures (clinical presentation, radiology, microbiology, pathology, organ involvement); medical and surgical treatment (including prior exposure to antifungals); response to treatment (clinical and radiological) at day 14, 42, 84; overall survival at day 14, 42, 84 and at last contact; and cause of death (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients diagnosed with an IA in 2016 and later
* Patients with a hematological malignancy
* Evidence of invasive Aspergillosis
* Aspergillus fumigatus culture from clinical material of the patient

Exclusion Criteria:

* Colonization only, without proof of invasive infection
* Non-availability of the azole resistant isolate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases will be recruited worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Treatment response to antifungal therapy in patients with an invasive Aspergillosis caused by an azole resistant pathogen. | Change from diagnosis at day 14, 28, 42 and 84 and throughout study completion
  Analysis of efficacy of antifungal therapy of azole-resistant and azole-susceptible invasive Aspergillosis. Patient receive either complete response, partial response, stable disease, progression of the disease. Treatment response will be assessed by treating physicians. Response will be compared between the two groups.

SECONDARY OUTCOMES:
Overall survival | 4 years
  Final outcome will be compared between the two groups in consideration of the type and state of underlying diseases and risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A. Cornely, Prof., Principal Investigator — University Hospital of Cologne, Germany; Paul E. Verweij, Prof., Principal Investigator — Radboud University Nijmegen Medical Center, The Netherlands
Locations (2):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with unauthorized persons. Anonymized data will only be exchanged between study coordinators and the analysis team.